CLINICAL TRIAL: NCT01070199
Title: Effects of Food Form and Fitness on Appetite and Digestion.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Purdue University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Richard Mattes, PhD, Purdue University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: R01DK079913 (NIH); R01DK079913 (NIH); 0805006922 (Other: Purdue University)
Record Dates: First submitted 2010-02-16; First posted 2010-02-17 (Estimated); Last update posted 2011-07-25 (Estimated); Status verified 2011-07

CONDITIONS: High and Increasing Contribution of Energy From Beverages in the Diet May Enhance Positive Energy Balance and Weight Gain
Keywords: obese, liquid, solid, fitness, humans, appetite
MeSH Terms: conditions — Weight Gain; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- liquid to liquid, (Experimental)
  Interventions: Behavioral: liquid to liquid
- liquid to solid, (Experimental)
  Interventions: Behavioral: liquid to solid
- solid to liquid (Experimental)
  Interventions: Behavioral: solid to liquid
- solid to solid (Experimental)
  Interventions: Behavioral: solid to solid

INTERVENTIONS:
Behavioral: liquid to liquid — • One test session will involve presentation of a glass of clear cherry-flavored unthickened beverage (Kool-Aid, Kraft Foods Inc., White Plains, NY). This session will be referred to as the "Liquid to Liquid" session as the participants will be consuming a liquid and be told that the consistency in their stomach will be a liquid.
  Other Names: Liquid test load
  Arms: liquid to liquid,
Behavioral: liquid to solid — This session involves a solution of calcium chloride and a solution of sodium alginate. The participant will be instructed to pour the cherry-flavored beverage/alginate solution into the calcium chloride. The result is a solid mass. They are allowed to examine the solution to confirm the solid texture and consistency.Participants will be told that this same reaction will occur in their stomach when the session's beverage is consumed due to the effect of gastric acid on the solution. But, the participant will be consuming the same cherry-flavored beverage as in the 1st session. Thus, they will believe that their GI tract will be challenged with a solid mass, but in reality, the challenge is the same (i.e., liquid).Therefore, the only difference between the test sessions is expectation.
  Other Names: liquid test load
  Arms: liquid to solid,
Behavioral: solid to liquid — • This session will involve the same dense gelatin cubes previously described, but participants will be told that the solid cubes will turn to liquid when they come into contact with the acid in their stomach. This trial will be known as "Solid to Liquid". A demonstration of the "Solid to Solid" and "Solid to Liquid" phases will be shown to the participant before they consume the load. Both phases exhibited by placing two cubes into separate containers filled with similar looking clear liquids. The "Solid to Solid" phase container will contain cold water so the cube stays in solid form. The "Solid to Liquid" phase container will contain hot water that will quickly dissolve the cube into a liquid form.
  Other Names: liquid test load
  Arms: solid to liquid
Behavioral: solid to solid — Participants will be presented with dense gelatin cubes. These 1" x 1" x 1" cubes will have a solid appearance and require mastication, but is isocaloric to the beverage. However, after mastication and gastric processing, the solid rapidly breaks down into a clear fluid.However, participants will be informed that the cubes will remain the same solid consistency in their stomach. The masticatory process and stimulus form will be standardized through the use of a metronome. Participants will be required to chew the solid cube at a fixed rate prior to swallowing. Thus, adding to the cognitive impression that they are eating a solid when essentially the GI challenge will be similar to the beverage.
  Other Names: liquid test load
  Arms: solid to solid

SUMMARY:
Energy-yielding fluids induce weaker appetitive and compensatory dietary responses than energy-matched semi-solids or solids. This is problematic because the high and increasing contribution of energy from beverages in the diet may enhance positive energy balance and weight gain. The prevailing view of the overweight/obesity problem is that it stems from a small, sustained positive energy balance. It follows then that only small changes, perhaps manipulations in the rheological characteristics of the diet, will be required to correct the problem. Certain populations that are more prone to weight gain may benefit from such manipulations. Obese individuals have a higher beverage intake and experience greater weight loss with reductions in beverage intake. Further, there is evidence that obese individuals consume more energy after a liquid pre-load than their lean counterparts, yet there is no difference in energy intake after a solid load. In contrast, habitual exercisers have been shown to have an increased accuracy of short-term regulation of food intake at meals following liquid preloads. A better understanding of the mechanisms by which beverages and energy-matched solid food forms elicit differential appetitive and dietary responses in these populations needed. This research will attempt to identify the influence of physical fitness and body fat on the ability to compensate for the energy content of solid and liquid preloads by reduction in energy intake at a subsequent ad libitum meal (i.e., acute compensation) and over the course of the day (i.e., short-term compensation). Furthermore, this study will examine the cognitive contribution to differential responses to energy-matched beverage and solid food forms and the effects of mastication on appetite, GI transit, glycemic response, and selected endocrine responses.

ELIGIBILITY:
Inclusion Criteria:

* 18-50 years of age BMI of 18-23 kg/m2 (lean) or 30-35 kg/m2 (obese) Sedentary physical activity level (<70th¬ percentile of estimated VO2max for age and sex) or physically Active/Exercisers (>70th¬ percentile of estimated VO2max for age and sex) Good health and not taking any medications known to influence appetite Non-smokers Not pregnant or lactating Weight stable (≤ 3 kg within last 3 months) Dietary restraint score <11 on the Three Factor Eating Questionnaire (included in the on-line screening questionnaire) Glucose Tolerant or Non-Diabetic (fasting blood glucose of <100 mg/dL) Self-reported consumer of breakfast and lunch

Exclusion Criteria:

* History or presence of significant metabolic diseases that may impact study results (i.e., endocrine, hepatic, renal disease) Individuals planning on starting a new diet or exercise regimen during the course of the study Use of obesity pharmacotherapeutic agents or over-the counter anti-obesity agents within the last 3 months Underlying conditions such as any cardiovascular, pulmonary, or neurological dysfunction that may be aggravated with exercise

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 81 (Actual)
Dates: Start 2009-01; Primary Completion 2009-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Change of energy intake. | 24 hours
  Effects of actual and perceived food form on short term energy intake in lean and obese, fit and unfit adults.

SECONDARY OUTCOMES:
Change of appetite. | 4 hours
  Effects of actual and perceived food form on hunger, fullness, desire to eat, and thirst.
Gastric emptying | 4 hours
  Effects of actual and perceived food form on gastric emptying time.
Gastro-intestinal transit | 4 hours
  Effects of actual and perceived food form on gastro-intestinal transit time.
Endocrin responses | 4 hours
  Effects of actual and perceived food form on GLP-1, CCK, Insulin, Ghrelin concentration.
Glucose response | 4 hours
  Effects of actual and perceived food form on serum glucose concentration.

CONTACTS AND LOCATIONS:
Locations (1):
- Purdue University, West Lafayette, Indiana, United States

REFERENCES:
- [Derived] Cassady BA, Considine RV, Mattes RD. Beverage consumption, appetite, and energy intake: what did you expect? Am J Clin Nutr. 2012 Mar;95(3):587-93. doi: 10.3945/ajcn.111.025437. Epub 2012 Jan 18. PMID 22258267